CLINICAL TRIAL: NCT05893342
Title: Perioperative Frailty and Postoperative Complications: a Prospective Study
Brief Title: Frailty in the Perioperative Period
Acronym: Frail-Negrin
Status: Recruiting | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Ángel Becerra-Bolaños, MD PhD, Principal Investigator, Dr. Negrin University Hospital
Other Study IDs: 2019-343-1
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Frailty
Keywords: Preoperative frailty; Postoperative complications
MeSH Terms: conditions — Frailty; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Preoperative frailty diagnostic — The preoperative evaluation of the patient will be carried out through the application of different scales that evaluate frailty (Edmonton frailty test, Barthel Index, Mini-mental test, Charlson Index) and a postoperative follow-up will be carried out for the diagnosis of complications during the first 90 postoperative days.

SUMMARY:
The presence of frailty is associated with a high risk of complications in the perioperative period, increasing morbidity and mortality, hospital stay, and loss of quality of life. In this prospective observational study, an evaluation of frailty was performed in patients older than 65 years old who undergo scheduled and urgent surgery. 138 patients are being included. The main objective is to evaluate the prevalence of frailty in patients older than 65 years undergoing surgery in our hospital and its association with postoperative mortality.

DETAILED DESCRIPTION:
The presence of frailty is associated with a high risk of complications in the perioperative period, increasing morbidity and mortality, hospital stay, and loss of quality of life. This is a prospective observational study in which an evaluation of frailty was performed in patients older than 65 years old who undergo scheduled and urgent surgery, including 138 patients. The main objective is to evaluate the prevalence of frailty in patients older than 65 years undergoing surgery and its association with postoperative mortality. The secondary objectives were the following: to assess the association between frailty and increased days of hospital stay, hospital readmission, and unexpected admission to ICU areas; to assess whether patients with greater frailty suffer a greater loss of postoperative functional independence; to evaluate type and frequency of complications; and to evaluate which scale is most useful to implement in the perioperative setting (Frailty Clinical Scale, Edmonton frailty test, Barthel Index, Mini-mental test, Charlson Index). Considering that the estimated percentage of frailty is 10%, with a 95% confidence interval and a 5% error margin, 138 patients are needed to accurately estimate the prevalence of frailty in the population.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years old undergoing urgent or scheduled surgery

Exclusion Criteria:

* Language barrier
* Cognitive impairment or inability to assist in clinical assessment during the study
* Refusal to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients over 65 years old undergoing surgery will be visited 24 hours before the intervention to sign the informed consent and the preoperative evaluation will be carried out through the application of different scales that evaluate the frailty of the patient. The patient will be monitored from his admission to the hospital until discharge and up to 3 months after the day of surgery. Data will be collected on in-hospital complications (medical or surgical), days of hospital stay, unforeseen need for ICU admission, if there has been loss of instrumental or cognitive abilities, and in-hospital mortality data and up to 3 months after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of frailty | First preoperative day
  Prevalence of frailty in patients older than 65 years undergoing surgery in our hospital
Postoperative complications | 90 postoperative days
  Relationship of preoperative frailty in patients older than 65 years undergoing surgery in our hospital and postoperative mortality

SECONDARY OUTCOMES:
Postoperative evolution | 90 postoperative days
  To evaluate the association between frailty and increased days of hospitalization, hospital readmission and unexpected admission to ICU areas.
Functional independence | First postoperative year
  To assess whether patients with greater frailty suffer a greater loss of postoperative functional independence.

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Becerra, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Doctor Negrín
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data could be available after request to the principal investigator